CLINICAL TRIAL: NCT04268329
Title: Evaluating the Use of an Informational Head and Neck Cancer Website for Patient and Family Education
Brief Title: Evaluating the Use of an Informational Head and Neck Cancer Website.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was not providing useful information.
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Virginie Achim, Assitant Professor, University of Illinois at Chicago
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-0725
Record Dates: First submitted 2020-01-30; First posted 2020-02-13 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: Patient's with head and neck cancer and 1 of their family members will be asked to visit an instructional head and neck cancer website to learn about what they might expect during the process of head and neck cancer treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational website: Patient (Other): Patients with a head and neck cancer will be asked to complete an 8 item questionnaire during their clinic visit. Patients will be shown the head and neck website (available in both English and Spanish) by a member of the study investigation team on a computer and also given the URL address to the study website. Patients will be asked to review the material on the website between their initial visit and there second follow-up visit. The time between visits will be between 1 and 4 weeks. Patients will be asked to record the number of times they visit the website and the time spent during each visit. Patients will be given a log sheet to document their use/time on the website. During the 2nd clinic visit patients will be asked to complete the same questionnaire that they completed during their initial study visit along with an additional 7 item survey. Following completion of the 2 documents, the patient's participation in the study will be completed.
  Interventions: Other: Educational website
- Educational website: Family member (Other): A family member of a patient with a head and neck cancer will be asked to complete an 8 item questionnaire during their clinic visit. They will be shown the head and neck website (available in both English and Spanish) by a member of the study investigation team on a computer and also given the URL address to the study website. They will be asked to review the material on the website between their relatives initial visit and there second follow-up visit. The time between visits will be between 1 and 4 weeks. The family member will be asked to record the number of times they visit the website and the time spent during each visit. They will be given a log sheet to document their use/time on the website. During the 2nd clinic visit the family member will be asked to complete the same questionnaire that they completed during their initial study visit along with an additional 7 item survey. Following completion of the 2 documents, their participation in the study will be completed.
  Interventions: Other: Educational website

INTERVENTIONS:
Other: Educational website — A website is used to educate patients and family members about head and neck cancer.
  Other Names: Educational Website: Patient; Educational Website: Family Member

SUMMARY:
It can be difficult for head and neck cancer patients and their families to fully understand the impact that cancer procedures and treatments can have on the cancer patients life. Procedures used to treat head and neck cancer may result in significant changes to the patients' physical appearance and/or functional abilities (talking, eating, and breathing). The lack of understanding as it relates to the effects of cancer treatments can have a significant impact on the patients post-operative success.

In an effort to help educate head and neck cancer patients and their families during this difficult time, the UIC department of Otolaryngology-HNS has created an informational website. The website is designed to educate cancer patients and their families regarding various cancer treatments and therapies.

DETAILED DESCRIPTION:
Head and neck cancer patients and their families often struggle to fully understand the degree to which cancer procedures and treatments may have on the cancer patient's life. The procedures involved in cancer treatment may result in significant changes to the patient's physical appearance and/or functional abilities (talking, eating, and breathing). Unfortunately, healthcare workers have a limited amount of time to spend educating their patients on all of the possibilities that may result from cancer related treatments. This lack of patient education and understanding can increase patient anxiety, compromise patient compliance, and result in less than optimum long-term outcomes.

Many patients are using the internet to educate themselves and to help them make their health care related decisions. However, for head and neck cancer patients, the information available on head and neck cancer websites is somewhat limited. In many cases, the information fails to provide adequate details as to the life changing, and at times disfiguring, results that head and neck cancer related treatments can have.

In an effort to help educate head and neck cancer patients and their families during this difficult time, the UIC department of Otolaryngology-HNS has created an informational website. The website includes information and educational videos about what to expect during the cancer treatment process. Specifically, the website is designed to educate cancer patients and their families on 1) the procedures that may be used to treat their specific cancer, 2) the side effects and post-operative hospital care of various treatments, 3) the physical changes that are possible as a result of their treatment, 4) functional changes that may occur as a result of their surgery/treatment, and 5) potential therapies that can be used to help improve their long-term outcome. The purpose of the website is to provide an educational and informative format, centered on head and neck cancer patients, that will help improve patient knowledge, understanding, and expectations during the course of cancer treatment and recovery.

Currently there are no studies that evaluate and or measure a change in patient/family member knowledge about head and neck cancer surgeries based on internet based information. However, there has been significant research related to the increased use of the internet for health care related decisions. These studies show that patients and families are more frequently turning to the internet and other forms of social media to learn about their diagnosis in order to make informed decisions about their medical care. Studies have also shown that websites are often written at a level well above the recommended reading level thereby inhibiting patient education.

3.0 Objectives/Aims

The objectives of this research are to evaluate 1) the change in subject knowledge before and after using the study head and neck cancer website, and 2) to determine whether a head and neck website is beneficial to study subjects in providing information that will result in improved compliance and ultimately long-term outcomes. Specifically, the PI's will be evaluating how the website educates cancer patients and their families on 1) the procedures that may be used to treat their specific cancer, 2) the side effects and post-operative care of various treatments, 3) the physical changes that are possible as a result of their treatment, 4) functional changes that may occur as a result of their surgery/treatment, and 5) potential therapies that can be used to minimize the physical and functional changes that may result from their cancer care.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects greater than 18 years of age.
2. Subjects that present to the UIC dept. of Otolaryngology-HNS with a head and neck cancer requiring surgery of the tongue, mandibulectomy, neck dissection, laryngectomy, or tracheostomy surgery and that have not previously had head and neck cancer resection surgery. (The surgeries listed are currently available on the website.)
3. One (1) family member of the cancer subject who will be treated at UIC for a head and neck cancer as noted in item 2 above, and who have not had a head and neck cancer surgery resection themselves. Patients undergoing treatment will remain eligible to participate independent of whether or not their family member takes part in the study.
4. Subjects that have access to the internet to view the study website either by using a desktop or laptop computer, a tablet or a smartphone.
5. Subjects who are willing to document their time on the website for study purposes.
6. Both English and Spanish speaking subjects who are literate and are able to read from a computer screen.
7. Subjects that understand the purpose and procedures of the study, who wish to participate, and who sign the study consent.

Exclusion Criteria:

1. Subjects under 18 years of age.
2. Subjects who do not have a head and neck cancer, or a family member with recently diagnosed head and neck cancer, or who have already had a head and neck cancer resection surgery.
3. Subjects that do not have access to the internet.
4. Subjects that do not understand or are not willing to follow the procedures as outlined in the study consent.
5. Subjects and/or their family member who cannot read or are legally blind.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-08-16 (Actual); Primary Completion 2020-06-18 (Actual); Study Completion 2020-06-18 (Actual)

PRIMARY OUTCOMES:
Evaluating the change in knowledge of head and neck cancer procedures before and after participants use of the study head and neck cancer website. | 4 weeks
  Participants will be asked to complete an 8 item questionnaire measurement tool (Website Study Questionnaire) about head and neck cancer procedures during their initial study visit. The questionnaire will be used to measure the participant's understanding of head and neck procedures before and after the use of an educational website. The participants will be provided a link to an educational website about head and neck cancer and they will be asked to view the website on several occasions in order to learn more about head and neck cancer procedures and what they or their family member might experience during and after their treatments. One to 4 weeks after the initial visit the participant will be asked to once again complete the same 8 item questionnaire. An increase in knowledge will be measured by counting the number of correct answers on the questionnaires before and after use of the website.

SECONDARY OUTCOMES:
The correlation between the use of an instructional head and neck cancer website and knowledge about head and neck cancer as measured by a study questionnaire. | 4 weeks
  Participants will be asked to record the time and date they visit the website onto a provided study log sheet. The number of correct answers recorded by participants during the completion of the second visit questionnaire will be correlated to the amount of time the participant spent using the educational website. It is expected that participants that visit and spend the greatest amount of time reviewing the website will have a greater understanding (a better questionnaire score) than participants that fail to use the website or who use of the website minimally.
  Participants will also complete an Otolaryngology/Head and Neck Surgery Website Study Survey that will be used to qualitatively measure if the participant found the educational website to be useful in their understanding of head and neck cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Virginie Achim, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Case Report Forms (CRF), questionnaires, and surveys will be assigned a code number that corresponds to the participant. A copy of the master list with subject name, MRN, and code number will be maintained by the study investigator in a separate file on a secured, password protected, encrypted UI Health System server. The coded data, without PHI, will be maintained on study personnel laptop computers. A hard copy of each subject's consent will be kept by the PI in a locked office in the EEI clinic Rm 3.87.
  Study data will be gathered from the cancer subjects medical record, directly from study subjects, and from completed surveys and questionnaires. Data with the linking code for each subject will be kept in an excel file database on an encrypted password protected laptop computer. Only approved study personnel will have access to the study data and the Master List.

REFERENCES:
- [Background] Kasabwala K, Agarwal N, Hansberry DR, Baredes S, Eloy JA. Readability assessment of patient education materials from the American Academy of Otolaryngology--Head and Neck Surgery Foundation. Otolaryngol Head Neck Surg. 2012 Sep;147(3):466-71. doi: 10.1177/0194599812442783. Epub 2012 Apr 3. PMID 22473833
- [Background] Lopez-Jornet P, Camacho-Alonso F. The quality of internet sites providing information relating to oral cancer. Oral Oncol. 2009 Sep;45(9):e95-8. doi: 10.1016/j.oraloncology.2009.03.017. Epub 2009 May 19. PMID 19457707
- [Background] Rice RE. Influences, usage, and outcomes of Internet health information searching: multivariate results from the Pew surveys. Int J Med Inform. 2006 Jan;75(1):8-28. doi: 10.1016/j.ijmedinf.2005.07.032. Epub 2005 Aug 24. PMID 16125453